CLINICAL TRIAL: NCT01726322
Title: A Study to Determine Alteration of Hormone Levels in Premenopausal Patients Receiving Adjuvant or Neo-adjuvant Chemotherapy for Breast Cancer
Brief Title: Ovarian Reserve in Premenopausal Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: As per the HRBs new funding model, HRBs investment will not support costs associated with routine patient care or translational studies, biobanks, patient registries and questionnaires. Therefore, a decision was made to cease further study follow up.
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: CTRIAL-IE (ICORG) 10-16
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Premenopausal Breast Cancer; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, salivary samples and hair samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a translational, mutlicentre study. The aim of this study is to determine whether pre-treatment levels of hormones predict ovarian follicular reserve post adjuvant or neoadjuvant chemotherapy for breast cancer and chemotherapy induced amenorrhea.

DETAILED DESCRIPTION:
It is proposed that levels of AMH and inhibin A and B measured will give an indication of the residual ovarian reserve in women with breast cancer treated with chemotherapy. In addition, AMH might give an indication of the possible efficacy of GNRH agonists in fertility preservation and the effect on ovarian follicular reserve using different adjuvant chemotherapy regimens. Those likely to be offered GNRH agonists are younger women with no children and a wish to have some in the future. Older women who have completed their families are less likely to be offered a GNRH agonist.

ELIGIBILITY:
Inclusion Criteria:

1. Documented histological diagnosis of invasive breast cancer
2. Patient due to be treated with chemotherapy (neoadjuvant or adjuvant)*
3. Female patients aged between 18 and 50 years
4. Premenopausal status as defined by a hormone profile within the pre-menopausal range as defined by local lab

   OR The patient's last menstrual period had to be within the last 180 days

   OR An IUD is used for contraception.
5. Ability to provide written informed consent

   * Patients treated with GNRH agonist or adjuvant Herceptin or participating in other clinical trials are also eligible

Exclusion Criteria:

1. Patients with hypothalamic/pituitary disorder
2. History of ovarian tumour
3. Current pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Premenopausal breast cancer patients who are to receive chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Alteration of hormone levels in premenopausal patients receiving adjuvant or neo-adjuvant chemotherapy for breast cancer | AMH levels will be taken at specified intervals until 3 years post chemotherapy
  To determine alteration of hormone levels in premenopausal patients receiving adjuvant or neo-adjuvant chemotherapy for breast cancer

SECONDARY OUTCOMES:
Comparative ovarian toxicity of differing neo-adjuvant/ adjuvant chemotherapy regimens | up to 3 years post chemotherapy
  To evaluate the comparative ovarian toxicity of differing neo-adjuvant/ adjuvant chemotherapy regimens
Correlation between CIA and depletion of ovarian follicular reserve. | up to 3 years post chemotherapy
  To assess the correlation between CIA and depletion of ovarian follicular reserve.
Correlation between changes in hormone levels during chemotherapy and the quality of life of premenopausal breast cancer patients | up to 3 years post chemotherapy
  To determine the correlation between changes in hormone levels during chemotherapy and the quality of life of premenopausal breast cancer patients
Efficacy of GNRH agonists in preservation of ovarian follicles in premenopausal women treated with adjuvant or neo-adjuvant chemotherapy for breast cancer | up to 3 years post chemotherapy
  To determine the efficacy of GNRH agonists in preservation of ovarian follicles in premenopausal women treated with adjuvant or neo-adjuvant chemotherapy for breast cancer (administration of GNRH agonists is dependent on the treating oncologist's judgment of the patient's case and prac-tices and is not to be influenced by study participation).

CONTACTS AND LOCATIONS:
Locations (10):
- Ireland (10):
  - Beacon Hospital, Dublin, Dublin 18
  - Our Lady of Lourdes Hospital, Drogheda, Louth
  - Bon Secours Hospital, Cork
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St James Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - Tallaght University Hospital, Dublin
  - Sligo General Hospital, Sligo
  - Waterford Regional Hospital, Waterford